CLINICAL TRIAL: NCT00187356
Title: Multicentre Radial Artery Patency Study: Results of Patency Beyond 5 Years After Coronary Artery Bypass Surgery
Acronym: RAPS - 5 years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Stephen E. Fremes, Head, Division of Cardiac and Vascular Surgery and Dr. Bernard S. Goldman Chair in Cardiovascular Surgery, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIHR MCT# 52681
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Bypass Surgery; Coronary Artery Disease; Angiography; Arterial Grafts; Radial Artery; Saphenous Vein
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- Surgical Conduit (Experimental): The surgical arm will be composed of the experimental arm (the use of the radial artery) versus an active comparator (the use of the saphenous vein graft).
  Interventions: Procedure: Radial Artery and Saphenous Vein Grafts Randomized to either right coronary or left circumflex coronary artery territories

INTERVENTIONS:
Procedure: Radial Artery and Saphenous Vein Grafts Randomized to either right coronary or left circumflex coronary artery territories — Each patient will receive both study grafts (Radial artery and Study Saphenous vein graft). The within-patient randomization scheme will dictate whether the radial goes to the right or circumflex territory. The saphenous vein graft will go to the opposing territory.

SUMMARY:
Bypass surgery is often required to treat severe coronary heart disease. Either arteries or veins can be used as bypass grafts. We wish to compare the long-term durability of the saphenous vein from the leg to that of the radial artery from the fore-arm when used as bypass grafts. We are examining how many of these grafts are still functioning beyond 5 years after bypass surgery by performing a coronary angiogram. After 1-year, we found that radial arteries were more likely to be functioning than saphenous veins. We hypothesize that radial arteries will continue to be superior beyond 5 years.

DETAILED DESCRIPTION:
The multi-centre Radial Artery Patency Study, (RAPS) is a series of longitudinal graft patency studies designed to compare the long-term patency of the radial artery to the saphenous vein. Between 1996 and 2001, 561 patients were intraoperatively randomized to undergo surgery according to one of two strategies: radial-artery grafting to the circumflex territory and saphenous-vein grafting to the right coronary artery or radial-artery grafting to the right coronary artery and saphenous-vein grafting to the circumflex territory. The first study compared the 8-12 month angiographic patency of the radial artery with that of the saphenous vein as a conduit for coronary artery bypass and found that radial arteries were superior. The primary objective of this current study is to determine the beyond 5-year angiographic patency of the radial artery compared with a saphenous vein coronary bypass graft.

HYPOTHESES

1. The angiographic patency of radial artery grafts studied beyond 5 years following surgery exceeds that of saphenous vein grafts.
2. Radial artery conduits studied beyond 5 years postoperatively have less graft disease than saphenous veins.

SAMPLE SIZE We expect to study 350 patients, which will allow us to test for a 35% risk reduction from 23% occlusion rate in saphenous veins to 15% in radial arteries, assuming a 5% within-patient correlation, with 80% power for a 2-tailed alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

The patient population consists of patients who were enroled into the original Multicentre Radial Artery Patency Study between November 1996 and January 2001. These included patients undergoing isolated coronary artery bypass surgery less than 80 years of age with 3 vessel coronary disease and left ventricular ejection fraction greater than 35%.

Exclusion Criteria:

Exclusion criteria included 1: Inability to use the radial artery or saphenous vein conduits: a)nonpalpable ulnar arteries or a positive Allen's test, b) an abnormal Doppler study or ultrasonographic study of the arms, c) a history of vasculitis or Raynaud's syndrome, bilateral varicose veins or vein stripping. 2: Conditions that affected the safety of follow-up angiography: a)renal insufficiency (creatinine > 180 umol/L) b)severe peripheral vascular disease precluding femoral access b)coagulopathy or obligatory uninterrupted use of anticoagulants c) known allergy to radiographic contrast media d) women of childbearing potential e) comorbid illness which precludes the use of follow up angiography f) geographically inaccessible for follow up angiography.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2002-07; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the proportion of grafts which are functionally occluded (TIMI flow 0, 1, or 2). | Beyond 5 years after bypass urgery

SECONDARY OUTCOMES:
a) the proportion of occluded study grafts (TIMI 0) | Beyond 5 years after bypass urgery
b) the proportion of functionally occluded grafts where proximal stenosis of native vessel is <90% vs >90% | Beyond 5 years after bypass urgery
c) the proportion of completely occluded grafts where proximal stenosis of native vessel is <90% vs >90% | Beyond 5 years after bypass urgery
d) proportion of study grafts with string sign | Beyond 5 years after bypass urgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Fremes, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (13):
- Canada (12):
  - University of Alberta, Edmonton, Alberta
  - Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - London Health Sciences Centre - UC, London, Ontario
  - London Health Sciences Centre - VC, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook and Women's College HSC, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Vancouver General Hospital, Vancouver, Ontario
  - Laval Hospital, Laval, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Montreal Jewish General Hospital, Montreal, Quebec
- Waikato Hospital, Hamilton, New Zealand

REFERENCES:
- [Background] Fremes SE. Multicenter radial artery patency study (RAPS). Study design. Control Clin Trials. 2000 Aug;21(4):397-413. doi: 10.1016/s0197-2456(00)00059-3. PMID 10913815
- [Result] Desai ND, Cohen EA, Naylor CD, Fremes SE; Radial Artery Patency Study Investigators. A randomized comparison of radial-artery and saphenous-vein coronary bypass grafts. N Engl J Med. 2004 Nov 25;351(22):2302-9. doi: 10.1056/NEJMoa040982. PMID 15564545
- [Result] Deb S, Cohen EA, Singh SK, Une D, Laupacis A, Fremes SE; RAPS Investigators. Radial artery and saphenous vein patency more than 5 years after coronary artery bypass surgery: results from RAPS (Radial Artery Patency Study). J Am Coll Cardiol. 2012 Jul 3;60(1):28-35. doi: 10.1016/j.jacc.2012.03.037. PMID 22742399
- [Derived] Tam DY, Deb S, Nguyen B, Ko DT, Karkhanis R, Moussa F, Fremes J, Cohen EA, Radhakrishnan S, Fremes SE. The radial artery is protective in women and men following coronary artery bypass grafting-a substudy of the radial artery patency study. Ann Cardiothorac Surg. 2018 Jul;7(4):492-499. doi: 10.21037/acs.2018.05.19. PMID 30094213
- [Derived] Deb S, Singh SK, Moussa F, Tsubota H, Une D, Kiss A, Tomlinson G, Afshar M, Sless R, Cohen EA, Radhakrishnan S, Dubbin J, Schwartz L, Fremes SE; Radial Artery Patency Study Investigators. The long-term impact of diabetes on graft patency after coronary artery bypass grafting surgery: a substudy of the multicenter Radial Artery Patency Study. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1246-53; discussion 1253. doi: 10.1016/j.jtcvs.2014.06.057. Epub 2014 Jul 17. PMID 25109754
- [Derived] Yanagawa B, Algarni KD, Singh SK, Deb S, Vincent J, Elituv R, Desai ND, Rajamani K, McManus BM, Liu PP, Cohen EA, Radhakrishnan S, Dubbin JD, Schwartz L, Fremes SE. Clinical, biochemical, and genetic predictors of coronary artery bypass graft failure. J Thorac Cardiovasc Surg. 2014 Aug;148(2):515-520.e2. doi: 10.1016/j.jtcvs.2013.10.011. Epub 2013 Dec 9. PMID 24332189